CLINICAL TRIAL: NCT06472011
Title: Back to the Basics: Metabolic and Appetitive Characteristics of Meals
Brief Title: Effects of Common Meals on Appetite and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HS-2024-0114
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Cheese

STUDY DESIGN:
Intervention Model Description: 7 crossover arms for each subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm 1 (lean steak and potatoes) (Experimental): lean steak and potatoes will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: lean steak and potatoes
- Arm 2 (lentil and sweet potato chili ) (Experimental): lentil and sweet potato chili will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: lentil and sweet potato chili
- Arm 3 (macaroni and cheese) (Experimental): macaroni and cheese will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: macaroni and cheese
- Arm 4 (fish tacos) (Experimental): fish tacos will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: fish tacos
- Arm 5 (chicken and pea fried rice) (Experimental): chicken and pea fried rice will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: chicken and pea fried rice
- Arm 6 (pita and hummus) (Experimental): pita and hummus will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: pita and hummus
- Arm 7 (creamy pork pasta) (Experimental): creamy pork pasta will be provided to subjects and primary and secondary outcomes will be measured at timelines explained under primary and secondary outcome measures.
  Interventions: Other: creamy pork pasta

INTERVENTIONS:
Other: lean steak and potatoes — Participants will be fed ~400 kcal lean steak and potatoes on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 1 (lean steak and potatoes)
Other: lentil and sweet potato chili — Participants will be fed ~400 kcal lentil and sweet potato chili on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 2 (lentil and sweet potato chili )
Other: macaroni and cheese — Participants will be fed ~400 kcal macaroni and cheese on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 3 (macaroni and cheese)
Other: fish tacos — Participants will be fed ~400 kcal fish tacos on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 4 (fish tacos)
Other: chicken and pea fried rice — Participants will be fed ~400 kcal chicken and pea fried rice on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 5 (chicken and pea fried rice)
Other: pita and hummus — Participants will be fed ~400 kcal pita and hummus on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 6 (pita and hummus)
Other: creamy pork pasta — Participants will be fed ~400 kcal creamy pork pasta on one occasion to test for changes in blood glucose and insulin levels as well as appetite over a 4-hour period of time.
  Arms: Arm 7 (creamy pork pasta)

SUMMARY:
The objectives of this study are to assess the impacts of meals composed of lean steak and potatoes (with a small portion of broccoli) in comparison to other common entrée/starch food combinations on metabolic and appetite responses.

DETAILED DESCRIPTION:
The objectives of this study are to utilize a novel, ecologically sound approach to assess the acute impacts of meals composed of lean steak and potatoes to other common entrée/starch food/vegetable combinations on metabolic and appetitive responses. Appetitive responses will serve as the primary outcome. Combinations for comparison will include lentil and sweet potato chili, macaroni and cheese, fish tacos, chicken and pea fried rice, pita and hummus, and creamy pork pasta.

ELIGIBILITY:
Inclusion Criteria:

* ages of 18-50 years
* BMI between 18-26

Exclusion Criteria:

* special dietary needs (e.g., gluten-free, etc.),
* 5% weight change in the previous 2 months,
* smoking, and substance use.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
appetite response | baseline (B), 15 minutes from B, 30 minutes from B, 45 minutes from B, 60 minutes from B, 90 minutes from B, 120 minutes from B, 150 minutes from B, 180 minutes from B, 210 minutes from B, 240 minutes from B
  Using 100 mm visual analog scales (score from 0 to 100 and higher score means more)

SECONDARY OUTCOMES:
blood glucose | baseline (B), 15 minutes from B, 30 minutes from B, 45 minutes from B, 60 minutes from B, 90 minutes from B, 120 minutes from B, 150 minutes from B, 180 minutes from B, 210 minutes from B, 240 minutes from B
  measuring blood glucose level

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided